CLINICAL TRIAL: NCT06973694
Title: Validation of Bulbicam Used on Patient Suffering From Diabetes Without Retinopathy
Status: Completed | Type: Observational
Sponsor: Meddoc (Other)
Responsible Party: Principal Investigator, Prof Stig Larsen, Research Director, Meddoc
Other Study IDs: V4-OTH/D-I/2023
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Diabetes
Keywords: Bulbicam; Reliability; Stability; Validity
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Diabetic patients: Patients suffering from diabetes without retinopathy of both genders with various durations of disease
  Interventions: Device: Bulbicam
- Age-matched healthy controls: Age-matched healthy controls without any eye diseases except for mild catarakt.
  Interventions: Device: Bulbicam

INTERVENTIONS:
Device: Bulbicam — The multi-test device, BulbiCam (BCAM), is a combined eye tracking; pupil metric; video graphic dual device which include the following 10 tests under development and ready for validation:
  26 grids glaucoma screening perimetry 64 grids full perimetry (NeuroField64) Pupil and Relative Afferent Pupil Defect (RAPD) assessment Semi-automatic ptosis (droopy eyelid) grading Video-based nystagmus test Dynamic acuity and contrast sensitivity test Dark adaptation test Smooth pursuit eye movements Saccade movements Eye fixation stability BCAM is connected to the BulbiHub software where measured data is stored and presented in numbers, diagrams, and graphs.

SUMMARY:
- The study consists of the following two study populations: 1) Patients suffering from diabetes without retinopathy of both genders with various durations of disease 2) Age-matched healthy control (HC) without any eye diseases except for mild catarakt.

Six bulbicam tests together with the standard method will be used in the study.

* The study will be performed as a controlled, open, and non-randomized observational multicenter study. For each included patient and age-matched HC will be included. All included participants will perform Bulbicam eye-investigation six times within three flowing days with a rest period of at least one hour. Each investigation includes same six Bulbicam tests. The standard method will only be performed once as the first investigation at day 1.
* The main variables will be the variables recorded at the four ACOLAPT- and two Pupil Bulbicam tests.
* Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. The Bulbicam examination will be performed twice a day with a rest period of one hour between each registration. This procedure will be repeated the following two days. All demographic data, social factors and history of disease will be recorded at screening. Additionally, the quality of life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be recorded initially as individual baseline values.

The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for measuring and classifying the tolerability and toxicity at the end of each day of investigation.

- Sixteen diabetes-patients with eaual many age-matched HC will be included.

DETAILED DESCRIPTION:
* The study consists of the following two study populations: 1) Patients suffering from diabetes without retinopathy of both genders with various durations of disease 2) Age-matched healthy control (HC) without any eye diseases except for mild catarakt.
* The six bulbicam tests "Visual acuity", "Contrast sensitivity", "Light adaptation latency with fixed frequency and variable contrast", "Light adaptation latency with variable frequency and fixed contrast" and "two pupil tests will be used. The Standard Method will be used initially for measurements of "iCare", "Visual acuity", "Refraction", "Contrast", "OCT" and "Fundus photography".
* The study will be performed as a controlled, open, and non-randomized observational multicenter study. For each included patient and age-matched HC will be included. All included participants will perform Bulbicam eye-investigation six times within three flowing days with a rest period of at least one hour. Each investigation includes same six Bulbicam tests. The standard method will only be performed once as the first investigation at day 1
* The main variables will be the variables recorded at the four ACOLAPT- and two Pupil Bulbicam tests.
* Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. The Bulbicam examination will be performed twice a day with a rest period of one hour between each registration. This procedure will be repeated the following two days. All demographic data, social factors and history of disease will be recorded at screening. Additionally, the quality of life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be recorded initially as individual baseline values.

The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for measuring and classifying the tolerability and toxicity at the end of each day of investigation.

* Sixteen diabetes-patients with eaual many age-matched HC will be included.

ELIGIBILITY:
Inclusion Criteria:

* Consists of patients diagnosed with Diabetes without retinopathy of both gender; passed the age of 18 years without any other eye disease; suffering from other know serious disease.

but have a health situation in accordance with expectations related to the age.

* Gender- and age-matched controls to patients in, passed the age of 18 years without any eye diseases; not suffering from other know serious disease and have a health situation in accordance with expectations related to the age.

Exclusion Criteria:

* Other visual disturbances and blindness
* Posterior Chamber Intra Ocular Lens (PCIOL)
* Physical or psychiatric disease, which may disturb the measuring procedure
* Patients who are not able to perform eye movements, so no full paresis of any ocular muscles.
* Patients whose visual acuity is less more than 1 logMAR in any eye, as these will not be able to focus on the test stimuli.
* Patients whose visible part of the eye is abnormal, such as subconjunctival hemorrhages or deformed pupils.
* Patients whose pupils are not able to respond normally to dilation or contraction due to damaged nerves, mechanical damage of the pupil etc.
* Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
* With known alcoholic and drug dependency
* Not able to understand information.
* Not willing to give written consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of Diabetic patients without retinopathy and healthy controls fulfilling the inclusion criteria and avoiding the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
1.Acolapt | 0 hours
  logMAR
2.Acolapt | 2 hours
  logMAR
3. Acolapt | 3 hours
  logMAR
4. Acolapt | 4 hours
  logMAR
5. Acolapt | 5 hours
  logMAR
6. Acolapt | 6 hours
  logMAR

SECONDARY OUTCOMES:
7.Contrast sensitivity | 0 hours
  Pelli-Robson score
8.Contrast sensitivity | 2 hours
  Pelli-Robson score
9. Contrast sensitivity | 3 hours
  Pelli-Robson score
10. Contrast sensitivity | 4 hours
  Pelli-Robson score
11. Contrast sensitivity | 5 hours
  Pelli-Robson score
12. Contrast sensitivity | 6 hours
  Pelli-Robson score

CONTACTS AND LOCATIONS:
Overall Officials: Goran Petrovski, PhD, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway